CLINICAL TRIAL: NCT01783938
Title: An Open-Label, Randomized, Phase 2 Study of Nivolumab Given Sequentially With Ipilimumab in Subjects With Advanced or Metastatic Melanoma
Brief Title: Study of Nivolumab Given Sequentially With Ipilimumab in Subjects With Advanced or Metastatic Melanoma (CheckMate 064)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-064
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Results first posted 2016-04-11 (Estimated); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Advanced or Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A: Nivolumab followed by Ipilimumab (Experimental): Nivolumab 3 mg/kg solution intravenously every 2 weeks up to 6 doses in Induction period and 3 mg/kg solution intravenously every 2 weeks until disease progression, unacceptable toxicity, or withdrawal of consent in Continuation period for a maximum of 2 years from 1st study treatment in Induction Period 1.
  Ipilimumab 3 mg/kg solution intravenously every 3 weeks up to 4 doses in Induction period.
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Cohort B: Ipilimumab followed by Nivolumab (Experimental): Ipilimumab 3 mg/kg solution intravenously every 3 weeks up to 4 doses in Induction period.
  Nivolumab 3 mg/kg solution intravenously every 2 weeks up to 6 doses in Induction period and 3 mg/kg solution intravenously every 2 weeks until disease progression, unacceptable toxicity, or withdrawal of consent in Continuation period for a maximum of 2 years from 1st study treatment in Induction Period 1.
  Interventions: Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Nivolumab
  Other Names: BMS-936558
Biological: Ipilimumab
  Other Names: Yervoy

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a sequential combination therapy of Nivolumab and Ipilimumab

DETAILED DESCRIPTION:
In order to evaluate the potential synergistic activity of nivolumab and ipilimumab and also because there may be differences in biology between tumors which are stable or responding to therapy and those that are clinically progressing, this study, CA209064, looked at two sequential combination regimens in which the second agent is administered immediately after a pre-specified duration of therapy with the first agent and not delayed until the time of progression after the first agent. This sequential study design looked at pharmacodynamic changes during treatment with one agent which may predict clinical activity to subsequent treatment with the alternate agent. This was done because it has not been scientifically proven whether or not the order in which nivolumab and ipilimumab are given is clinically important.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histologically confirmed unresectable Stage III or IV melanoma
* Treatment-naive or experienced disease recurrence or progression during or after one prior systemic regimen for advanced disease
* Measurable disease by Computed Tomography/Magnetic resonance imaging (CT/MRI) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Known BRAF V600 mutation status or consent to BRAF V600 mutation testing
* Sufficient tumor tissue accessible for baseline and post-treatment biopsies.

Exclusion Criteria:

* Active central nervous system (CNS) metastases
* Carcinomatous meningitis
* Active, known or suspected autoimmune disease
* Condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization
* Prior therapy with anti-Programmed Death-1 (PD1), anti-Programmed Death-Ligand 1 (PD-L1), anti-PD-L2, anti-CD137, or anti-CTLA-4 (cytotoxic T lymphocyte antigen 4) antibody
* Prior treatment with other immunotherapies
* Prior therapy with BRAF inhibitor within 6 weeks of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2013-04-30 (Actual); Primary Completion 2015-04-03 (Actual); Study Completion 2020-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- United States (10):
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Indiana University Health Melvin And Bren Simon Cancer Center, Indianapolis, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University Of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- [Derived] Yoshida T, Ichikawa J, Giuroiu I, Laino AS, Hao Y, Krogsgaard M, Vassallo M, Woods DM, Stephen Hodi F, Weber J. C reactive protein impairs adaptive immunity in immune cells of patients with melanoma. J Immunother Cancer. 2020 Apr;8(1):e000234. doi: 10.1136/jitc-2019-000234. PMID 32303612
- [Derived] Weber JS, Gibney G, Sullivan RJ, Sosman JA, Slingluff CL Jr, Lawrence DP, Logan TF, Schuchter LM, Nair S, Fecher L, Buchbinder EI, Berghorn E, Ruisi M, Kong G, Jiang J, Horak C, Hodi FS. Sequential administration of nivolumab and ipilimumab with a planned switch in patients with advanced melanoma (CheckMate 064): an open-label, randomised, phase 2 trial. Lancet Oncol. 2016 Jul;17(7):943-955. doi: 10.1016/S1470-2045(16)30126-7. Epub 2016 Jun 4. PMID 27269740
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 140 randomized,138 treated because 1 experienced adverse event unrelated to study drug and 1 no longer met study criteria.
Groups:
- Nivolumab Followed by Ipilimumab: Nivolumab 3 mg/kg Q2W IV over 60 min for up to 6 doses during Weeks 1 to 13 in Induction Period 1 followed by Ipilimumab 3 mg/kg Q3W IV over 90 min for up to 4 doses during Weeks 13 to 25 in Induction Period 2.
- Ipilimumab Followed by Nivolumab: Ipilimumab 3 mg/kg Q3W IV over 90 min for up to 4 doses during Weeks 1 to 13 in Induction Period 1 followed by Nivolumab 3 mg/kg Q2W IV over 60 min for up to 6 doses during Weeks 13 to 25 in Induction Period 2.
Period: Overall Study
Arm/Group | Nivolumab Followed by Ipilimumab | Ipilimumab Followed by Nivolumab
Started | 68 | 70
Completed | 11 | 9
Not Completed | 57 | 61
Not completed — Disease Progression | 18 | 41
Not completed — Study Drug Toxicity | 27 | 14
Not completed — Adverse Event Unrelated to Study Drug | 4 | 2
Not completed — Participant Request to Discontinue Study Treatment | 2 | 3
Not completed — Participant Withdrew Consent | 2 | 0
Not completed — Maximum Clinical Benefit | 1 | 0
Not completed — Other Reasons | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab Followed by Ipilimumab | Ipilimumab Followed by Nivolumab | Total
Number analyzed (Participants) | 68 | 70 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (14.08) | 60.6 (15.17) | 59.8 (14.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 46 | 46 | 92
Race/Ethnicity, Customized [Number; unit: participants]
  White | 65 | 66 | 131
  Black or African American | 1 | 2 | 3
  Asian | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Other | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Related Grade 3-5 Adverse Events (AEs) During the Induction Period (Period 1 and 2)
Description: The percentage of participants with treatment-related grade 3-5 adverse events (AEs) is defined as the number of participants who experienced at least 1 treatment related grade 3 - 5 adverse event (AE) per national cancer institute common terminology criteria for adverse events (NCI CTCAE v4.0, any preferred term) with an onset date after or on first day of Induction Period #1 and not later than discontinuation date from Induction Period #2, divided by the total number of treated participants.
  Adverse Event (AE) = any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may or may not have a causal relationship with treatment.
  Treatment-related = having certain, probable, possible, or missing relationship to study drug.
  Grade (Gr) 3=Severe Gr 4=Potentially Life-threatening or disabling Gr 5=Death
Time Frame: From Day 1 to up to Week 25
Population: All treated participants
Measure: Number; unit: Percentage of participants
Arm/Group | Nivolumab Followed by Ipilimumab | Ipilimumab Followed by Nivolumab
Number analyzed (Participants) | 68 | 70
Percentage of participants | 64.7 [37.6 to 62.4] | 51.4 [31.1 to 55.3]

2. Secondary Outcome: Investigator-Assessed Response Rate at Week 25
Description: Response rate is defined as the number of participants who have a complete response (CR) or partial response (PR) at Week 25 per modified RECIST 1.1 criteria, with confirmation on the scheduled scan at Week 33 (or any subsequent scan performed at least 4 weeks after the Week 25 scan), divided by the total number of treated participants. Results of the tumor assessment at Week 13 or any unscheduled tumor assessment obtained prior to Week 25, except for baseline/screening tumor assessment, were not considered in the assessment of response rate at Week 25.
Time Frame: Week 25
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab Followed by Ipilimumab | Ipilimumab Followed by Nivolumab
Number analyzed (Participants) | 68 | 70
Percentage of participants | 54.7 [40.0 to 68.4] | 30.4 [17.7 to 45.8]

3. Secondary Outcome: Investigator-Assessed Duration of Response (DOR)
Description: Duration of response (DOR) is defined as the time between the Week 25 date of response and the date of objectively documented disease progression as defined by modified RECIST 1.1 criteria or death, whichever occurs first. Median computed using Kaplan-Meier method.
Time Frame: From week 25 to up to date of disease progression or death (Up to 6 years)
Population: All treated participants with confirmed response at week 25
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nivolumab Followed by Ipilimumab | Ipilimumab Followed by Nivolumab
Number analyzed (Participants) | 29 | 14
months | NA [25.40 to NA] — Median and upper limit not reached because of too few events to evaluate | 57.66 [13.67 to NA] — Upper limit not reached because of too few events to evaluate

4. Secondary Outcome: Investigator-Assessed Rate of Progression
Description: Progression rate at a specific timepoint is defined as the number of participants who have Progressive Disease (PD) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 at that specific timepoint divided by the total number of treated participants. As specified by modified RECIST 1.1, the evaluation of PD at Week 13 and Week 25 used the baseline tumor assessment as reference. A participant who died without a reported prior progression was considered to have progressed on the date of death. Deaths before or at Week 13 are counted as progression outcome. Confidence interval is based on the Clopper and Pearson method.
Time Frame: Week 13 and Week 25
Population: All treated participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab Followed by Ipilimumab | Ipilimumab Followed by Nivolumab
Number analyzed (Participants) | 68 | 70
Percentage of participants
  Week 13 | 36.8 [25.4 to 49.3] | 62.9 [50.5 to 74.1]
  Week 25 | 36.8 [25.4 to 49.3] | 60.0 [47.6 to 71.5]

ADVERSE EVENTS:
Time Frame: From first dose to 100 days post last dose (Up to 6 years)
Arm/Group | Nivolumab Followed by Ipilimumab | Ipilimumab Followed by Nivolumab
All-Cause Mortality (participants affected / at risk) | 35/68 | 48/70
Serious Adverse Events (participants affected / at risk) | 59/68 | 57/70
Other Adverse Events (participants affected / at risk) | 68/68 | 68/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab Followed by Ipilimumab (N=68) | Ipilimumab Followed by Nivolumab (N=70)
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Addison's disease (Endocrine disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 5 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 1 | 2
Hypopituitarism (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Macular oedema (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 3
Autoimmune colitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 13 | 15
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 7
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 4
Pancreatitis acute (Gastrointestinal disorders) | 0 | 3
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Terminal ileitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 5
Asthenia (General disorders) | 0 | 3
Fatigue (General disorders) | 2 | 10
Gait disturbance (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 5 | 4
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hepatitis (Hepatobiliary disorders) | 3 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Autoimmune disorder (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Encephalitis (Infections and infestations) | 1 | 0
Infected cyst (Infections and infestations) | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 3
Sepsis (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 6
Wound infection (Infections and infestations) | 2 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 2
Hepatic enzyme increased (Investigations) | 1 | 0
Influenza A virus test positive (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 22
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Demyelinating polyneuropathy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Meningitis noninfective (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 5 | 3
Bladder spasm (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 2 | 1
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab Followed by Ipilimumab (N=68) | Ipilimumab Followed by Nivolumab (N=70)
Anaemia (Blood and lymphatic system disorders) | 25 | 25
Sinus tachycardia (Cardiac disorders) | 5 | 1
Adrenal insufficiency (Endocrine disorders) | 5 | 3
Hyperthyroidism (Endocrine disorders) | 3 | 4
Hypophysitis (Endocrine disorders) | 5 | 4
Hypothyroidism (Endocrine disorders) | 18 | 20
Diplopia (Eye disorders) | 1 | 4
Dry eye (Eye disorders) | 4 | 5
Photophobia (Eye disorders) | 4 | 1
Vision blurred (Eye disorders) | 10 | 10
Abdominal distension (Gastrointestinal disorders) | 5 | 5
Abdominal pain (Gastrointestinal disorders) | 17 | 24
Abdominal pain upper (Gastrointestinal disorders) | 5 | 6
Colitis (Gastrointestinal disorders) | 7 | 8
Constipation (Gastrointestinal disorders) | 27 | 30
Diarrhoea (Gastrointestinal disorders) | 44 | 38
Dry mouth (Gastrointestinal disorders) | 8 | 7
Dyspepsia (Gastrointestinal disorders) | 5 | 3
Dysphagia (Gastrointestinal disorders) | 4 | 4
Flatulence (Gastrointestinal disorders) | 3 | 7
Gastritis (Gastrointestinal disorders) | 4 | 2
Nausea (Gastrointestinal disorders) | 42 | 40
Vomiting (Gastrointestinal disorders) | 22 | 31
Asthenia (General disorders) | 4 | 6
Chills (General disorders) | 20 | 15
Fatigue (General disorders) | 56 | 59
Gait disturbance (General disorders) | 4 | 2
Influenza like illness (General disorders) | 12 | 1
Malaise (General disorders) | 3 | 6
Non-cardiac chest pain (General disorders) | 6 | 5
Oedema peripheral (General disorders) | 17 | 15
Pain (General disorders) | 6 | 8
Pyrexia (General disorders) | 30 | 22
Candida infection (Infections and infestations) | 2 | 6
Nasopharyngitis (Infections and infestations) | 6 | 5
Sinusitis (Infections and infestations) | 6 | 4
Skin infection (Infections and infestations) | 5 | 3
Upper respiratory tract infection (Infections and infestations) | 12 | 9
Urinary tract infection (Infections and infestations) | 9 | 8
Contusion (Injury, poisoning and procedural complications) | 4 | 6
Fall (Injury, poisoning and procedural complications) | 8 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 4
Alanine aminotransferase increased (Investigations) | 30 | 22
Amylase increased (Investigations) | 20 | 16
Aspartate aminotransferase increased (Investigations) | 28 | 22
Blood alkaline phosphatase increased (Investigations) | 17 | 14
Blood bilirubin increased (Investigations) | 10 | 3
Blood creatinine increased (Investigations) | 3 | 11
Blood thyroid stimulating hormone increased (Investigations) | 4 | 5
Blood urea increased (Investigations) | 4 | 3
Lipase increased (Investigations) | 28 | 23
Lymphocyte count decreased (Investigations) | 7 | 5
Platelet count decreased (Investigations) | 6 | 4
Weight decreased (Investigations) | 15 | 23
White blood cell count decreased (Investigations) | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 31 | 33
Dehydration (Metabolism and nutrition disorders) | 17 | 20
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 20 | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 12 | 10
Hypermagnesaemia (Metabolism and nutrition disorders) | 6 | 5
Hypernatraemia (Metabolism and nutrition disorders) | 4 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 16
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 24 | 21
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 22
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 21 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 | 7
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Dizziness (Nervous system disorders) | 18 | 10
Dysgeusia (Nervous system disorders) | 8 | 4
Headache (Nervous system disorders) | 31 | 17
Paraesthesia (Nervous system disorders) | 10 | 4
Anxiety (Psychiatric disorders) | 9 | 10
Confusional state (Psychiatric disorders) | 4 | 3
Depression (Psychiatric disorders) | 8 | 3
Insomnia (Psychiatric disorders) | 19 | 13
Haematuria (Renal and urinary disorders) | 6 | 3
Nocturia (Renal and urinary disorders) | 1 | 4
Pollakiuria (Renal and urinary disorders) | 4 | 4
Urinary tract pain (Renal and urinary disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 27
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 | 16
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 9
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 5 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 32 | 34
Rash (Skin and subcutaneous tissue disorders) | 32 | 25
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 17 | 15
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 7
Skin lesion (Skin and subcutaneous tissue disorders) | 4 | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 12 | 13
Hot flush (Vascular disorders) | 2 | 5
Hypertension (Vascular disorders) | 9 | 3
Hypotension (Vascular disorders) | 8 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2013-03-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT01783938/Prot_000.pdf
  • Statistical Analysis Plan (2014-03-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT01783938/SAP_001.pdf